CLINICAL TRIAL: NCT01505023
Title: Evaluation of the Effectiveness of a Partial Meal Replacement With Inulin on Obesity and Dyslipidemias in Women.
Brief Title: Partial Meal Replacement and Inulin in Obese Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cindetec (Other)
Collaborators: Nucitec SA de CV (Unknown)
Responsible Party: Principal Investigator, SANDRA GARCiA PADILLA, Clinical Research Coordinator, Cindetec
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEE-001-2004
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Partial meal replacement (Active Comparator)
  Interventions: Dietary Supplement: Partial meal replacement
- Partial meal replacement with inulin (Experimental)
  Interventions: Dietary Supplement: Partial meal replacement with inulin
- Inulin (Active Comparator)
  Interventions: Dietary Supplement: Inulin
- No intervention (No Intervention)

INTERVENTIONS:
Dietary Supplement: Partial meal replacement — The PMR was designed to contain sufficient amounts of all vitamins and minerals. Women were instructed to consume 2 servings per day at breakfast and dinner, each consisting of 33 g of powder dissolved in 250 ml of skim milk.
  Arms: Partial meal replacement
Dietary Supplement: Partial meal replacement with inulin — The PMR was designed to contain sufficient amounts of all vitamins and minerals plus inulin. Women were instructed to consume 2 servings per day at breakfast and dinner, each consisting of 33 g of powder dissolved in 250 ml of skim milk.
  Arms: Partial meal replacement with inulin
Dietary Supplement: Inulin — Women were asked to consume one 5g serving of inulin mixed with any drink at breakfast and same amount at dinner (10 g of inulin/d).
  Arms: Inulin

SUMMARY:
The objective of this study was to test the efficacy of a partial meal replacement added with vitamins, minerals and inulin on weight reduction, blood lipids and micronutrients intake in obese Mexican women

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m 2

Exclusion Criteria:

* Pregnant
* Lactating
* Diagnosed with diabetes
* Diagnosed with hypertension
* Fasting glucose ≥126 mg/dL
* Blood triglycerides ≥400mg/dL

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Weight
Blood lipids

SECONDARY OUTCOMES:
Micronutrients intake

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autónoma de Querétaro, Querétaro City, Querétaro, Mexico

REFERENCES:
- [Derived] Tovar AR, Caamano Mdel C, Garcia-Padilla S, Garcia OP, Duarte MA, Rosado JL. The inclusion of a partial meal replacement with or without inulin to a calorie restricted diet contributes to reach recommended intakes of micronutrients and decrease plasma triglycerides: a randomized clinical trial in obese Mexican women. Nutr J. 2012 Jun 18;11:44. doi: 10.1186/1475-2891-11-44. PMID 22703579